CLINICAL TRIAL: NCT04252638
Title: Acceptance and Commitment Therapy as a New Treatment for Adults With Insomnia Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-AI
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Insomnia Chronic
Keywords: Insomnia; Acceptance and Commitment Therapy; Cognitive Behavioral Therapy; Randomized Controlled Trial; Sleep; Quality of life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy plus Sleep Restriction (Experimental): Acceptance and Commitment therapy is a well-established treatment for other disorders including depression, anxiety and chronic pain, but has not been thoroughly investigated for insomnia. The therapy consists of mindfulness, acceptance, identification of personal life values and committed action. In addition, patients in this group will receive sleep restriction, a behavioral therapy component of cognitive behavioral therapy for insomnia. The treatment will consist of six weekly sessions of group psychotherapy and will be conducted in an outpatient setting.
  Interventions: Behavioral: Acceptance and Commitment Therapy plus Sleep Restriction
- Cognitive Behavioral Therapy including Sleep Restriction (Active Comparator): The control intervention is Cognitive Behavioral Therapy for insomnia (CBT-I). This is the first line treatment for adults with chronic insomnia. The therapy consists of education, relaxation, and behavioral therapy, including sleep restriction. The treatment will consist of six weekly sessions of group psychotherapy and will be conducted in an outpatient setting.
  Interventions: Behavioral: Cognitive Behavioral Therapy including Sleep Restriction

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy plus Sleep Restriction — Acceptance and Commitment Therapy (ACT) is a newer form of behavioral therapy working with acceptance, and the clarification of personal values. Acceptance, in this case, means the willingness to (temporarily) experience unpleasant sensations such as sleeplessness or tiredness without attempting to control or change them. Aims are, first, to reduce suffering due to unsuccessful control attempts (such as frustration, anger, anxiety) and second, to improve processes that are typically worsened by increased control efforts (such as sleep). Clarification of values means identifying aspects of life that are perceived as rewarding and encouraging approach-behavior in valued aspects of life (instead of avoidance-behavior that is often associated with insomnia and mental disorders).
  Arms: Acceptance and Commitment Therapy plus Sleep Restriction
Behavioral: Cognitive Behavioral Therapy including Sleep Restriction — CBT-I, the gold standard treatment for insomnia, consists of sleep education, relaxation, sleep restriction, and cognitive therapy.
  Arms: Cognitive Behavioral Therapy including Sleep Restriction

SUMMARY:
Acceptance and Commitment Therapy plus sleep restriction (ACT) will be compared to Cognitive Behavioral Therapy for insomnia (CBT-I). CBT-I is the first line treatment for insomnia according to current guidelines. The aim of the study is to investigate the efficacy of ACT, compared to CBT-I, for the improvement of sleep-related quality of life and insomnia severity.

DETAILED DESCRIPTION:
Insomnia is a major health problem worldwide and a risk factor for the onset of other diseases, including cardiovascular and mental disorders. The prevalence of insomnia is 10% in the adult population. Cognitive Behavioral Therapy for insomnia (CBT-I) is the most effective treatment according to current guidelines. However, with response rates of around 70% and remission rates of around 40%, many patients need additional treatment. Common difficulties are that i) behavioral treatment elements, especially sleep restriction, are not implemented by patients, and that ii) quality of life does not improve despite improvements in sleep. Long-term pharmacological treatment is not recommended because it is often associated with a loss of efficacy and the risk of severe side effects. The aim of this research project is to improve behavioral treatment options for patients with insomnia.

Acceptance and Commitment Therapy (ACT) is a new form of behavioral therapy. Efficacy, primarily an improvement of quality of life, has already been proven for other conditions including chronic pain and depression - however, no controlled study in patients with insomnia has yet been conducted. In a feasibility study, our workgroup provided first evidence that this treatment is feasible and potentially efficacious mainly for the improvement of sleep related quality of life. The current proposal is designed to extend this preliminary work in form of a prospective randomized controlled pilot trial. ACT will be compared with the gold standard treatment (CBT-I) in 60 patients with a primary diagnosis of insomnia disorder. The primary aim of this research is to test for differential efficacy, i.e. whether ACT is more effective for the improvement of i) insomnia severity and ii) sleep-related quality of life.

The planned study is prospective, randomized, controlled, confirmatory, two-armed, single-blinded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Ability to give written informed consent
* Sufficient fluency in German to participate in group therapy and fill in questionnaires
* Meeting research diagnostic criteria for insomnia disorder according to DSM 5

Exclusion Criteria:

* Serious medical condition (e.g. tumor disease, epilepsy, encephalitis, history of traumatic brain injury, other organic brain syndromes), severe heart disease and other debilitating or instable medical conditions or upcoming surgery
* Acute pain or poorly managed chronic pain
* Suicidality
* Severe psychiatric disorder (e.g. psychosis, bipolar disorder, borderline personality disorder, intellectual disability, autism) or other psychiatric disorder requiring treatment outside of study
* Alcohol or drug abuse or dependency including benzodiazepine dependency
* Evidence of untreated sleep apnea
* Evidence of restless legs syndrome
* Evidence of parasomnia
* Circadian rhythm disorder including night shift work
* Alteration of medication within 4 weeks prior to study treatment, stable medication does not lead to exclusion
* Current other psychotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Insomnia Severity at six weeks | change over six weeks (directly before and directly after therapy)
  The ISI is a valid, reliable and change-sensitive self-rating questionnaire that is widely used as an outcome measure in clinical trials in insomnia research. A self-rating questionnaire in contrast to objective sleep measures such as polysomnography or actigraphy is reasonable and widely accepted for measuring insomnia severity because insomnia is defined on the basis of subjective sleep perception and objective measures often deviate from this perception. Advantages of the ISI, compared to a sleep diary, are that it combines different aspects of insomnia such as sleep onset difficulties, sleep maintenance difficulties, and daytime impairment in one summary score, and that it is easier to use for patients. Following Morin et al., response is defined as an improvement of > seven points on the ISI. Remission is defined as a post-treatment ISI score of < 8. The minimum score is 0 points, the maximum score is 28 points. Higher score indicate more severe insomnia.
Change from Baseline Glasgow Sleep Impact Index at six weeks | change over six weeks (directly before and directly after therapy)
  In the GSII, patients are asked to specify the most important aspect of daytime functioning which they perceive to be negatively affected by their insomnia. The degree of impairment is rated on visual analogue scale. The minimum value of the scale is 0 points, the maximum value is 100 points. Higher values indicate better sleep-related quality of life.

SECONDARY OUTCOMES:
Change from Baseline Insomnia Severity at six months | change over six months (directly before therapy and six months later)
  The ISI is a valid, reliable and change-sensitive self-rating questionnaire that is widely used as an outcome measure in clinical trials in insomnia research. A self-rating questionnaire in contrast to objective sleep measures such as polysomnography or actigraphy is reasonable and widely accepted for measuring insomnia severity because insomnia is defined on the basis of subjective sleep perception and objective measures often deviate from this perception. Advantages of the ISI, compared to a sleep diary, are that it combines different aspects of insomnia such as sleep onset difficulties, sleep maintenance difficulties, and daytime impairment in one summary score, and that it is easier to use for patients. Following Morin et al., response is defined as an improvement of > seven points on the ISI. Remission is defined as a post-treatment ISI score of < 8. The minimum score is 0 points, the maximum score is 28 points. Higher score indicate more severe insomnia.
Change from Baseline Glasgow Sleep Impact Index at six months | change over six months (directly before therapy and six months later)
  In the GSII, patients are asked to specify the most important aspect of daytime functioning which they perceive to be negatively affected by their insomnia. The degree of impairment is rated on visual analogue scale. The minimum value of the scale is 0 points, the maximum value is 100 points. Higher values indicate better sleep-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Hertenstein, PhD, Principal Investigator — UPD Bern
Locations (1):
- Universitäre Psychiatrische Dienste Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No